CLINICAL TRIAL: NCT00617383
Title: Determine if the Presence of Characteristic MS-like Lesion(s) on Baseline MRI Predisposes to CIS/MS in Female MZ Twins Discordant for CIS/MS.
Brief Title: AT RISK FOR MS - Clinical Conversion of Female Monozygotic Twins Discordant for CIS/MS
Acronym: ARMS
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Other Study IDs: HSC-MS-07-0327; NMSS Pilot grant PP1464
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2012-02

CONDITIONS: Multiple Sclerosis; Clinically Isolated Syndrome
Keywords: demyelinating disease; multiple sclerosis; female monozygotic identical twins; MS; non-concordant; clinically isolated syndrome - CIS; brain MRI; proteomics
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood for serum and peripheral mononuclear cells; optional CSF - cerebrospinal fluid at entry and exit from trail
Oversight: Data Monitoring Committee: No

SUMMARY:
The definition of the most 'at-risk' population within highly susceptible groups would provide an opportunity for preemptive therapeutics.

A convenient, safe, and tolerable therapy that delays the onset of clinical disease during the pre-symptomatic stage of demyelinating disease would provide a therapeutic alternative to a 'wait and see' approach in subjects at 'high risk' for CIS (clinically isolated syndrome - monosymptomatic demyelinating disease) or MS.

Identical twins share the same genes and have the highest rate of shared MS. An identical female with a sister twin with MS has a 34% chance of having MS. Non concordant (no MS yet) identical (monozygotic - from the same sperm-egg zygote) female twins provide an ideal population to find out what factors predict the onset of MS in the non-affected twin.

We will recruit 30 identical female twins, one with MS and the other without MS, and obtain brain MRI and biological samples on the non-affected twin and determine if:

* the presence of characteristic MS-like lesion(s) on baseline MRI predisposes to MS.
* specific proteins in blood or cerebrospinal fluid predispose to the clinical expression of demyelinating disease

If we can predict by simple tests (MR brain scan and blood tests) the likelihood of the onset of MS in 'at risk' subjects, and have safe and tolerable therapies, we may be able to prevent the clinical onset of demyelinating disease (MS).

DETAILED DESCRIPTION:
Primary Objective: Determine if the presence of characteristic MS-like lesion(s) on baseline MRI predisposes to CIS/MS in female MZ twins discordant for CIS/MS.

Secondary Objective: Define the protein and microarray gene expression profile predictive of conversion to MS/CIS in female MZ twins discordant for CIS/MS.

Design and Outcomes: This is a single center, clinical study to determine if the presence of MS-like MRI brain lesions predict the rate of conversion to CIS in female MZ twins discordant for CIS/MS.

We will screen and recruit 30 subjects, and begin to follow these subjects annually for a total of 5 years to determine if MR brain scans predict CIS/MS conversion.

Interventions and Duration: Subjects will be recruited over 2 years and followed for five years with annual neurological examinations and MR brain scans.

Sample Size and Population: 30 female co-twins discordant for CIS/MS will be studied. We predict 72% of the 27% 'at risk' subjects with characteristic MR brain lesions at baseline will convert to CIS within 5 years. We predict only 6% of the 73% 'at risk' subjects without characteristic MR brain lesions at baseline will convert to CIS within 5 years.

These data will determine if paraclinical (MRI) evidence of demyelinating disease and specific blood or cerebrospinal fluid proteins predict clinical expression of disease in highly susceptible populations predicts.

ELIGIBILITY:
Inclusion Criteria:

* 'at risk' individuals for MS - female co-twins discordant for CIS/MS.
* 'at risk' individuals for MS who at the time of randomization have not converted to MS or CIS.
* 'at risk' individuals will be treatment-naïve for immunomodulatory/suppressive medications.
* < 46 years old.

Exclusion Criteria:

* Individuals diagnosed with MS or CIS.
* Other 'at risk' individuals who do not conform to the specific 'at risk' groups outlined above e.g., 1st degree, 2nd degree and 3rd degree relative of MS index cases.
* Subjects over 45.
* Use of immunomodulatory medications such as azathioprine, gold, sulfasalazine, minocycline, statins, and MTX or prednisone > 7.5 mg/day within 30 days of randomization for any reason.
* Active drug use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements or a psychiatric disorder that is unstable or would preclude reliable participation in the study.
* Serious illness (requiring systemic treatment and/or hospitalization) such as diabetes mellitus, renal, cardiac, or pulmonary disease. Subjects with a history of alcoholism, or in whom intellectual functioning is impaired sufficiently to interfere with the understanding of the protocol, or participation in the treatment and evaluation program.

Ages: 10 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: female monozygotic twins discordant for CIS/MS
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Determine if the presence of characteristic MS-like lesion(s) on baseline MRI predisposes to CIS/MS in female MZ twins discordant for CIS/MS. | 5 years or exit from study

SECONDARY OUTCOMES:
Define the protein and microarray gene expression profile predictive of conversion to MS/CIS in female MZ twins discordant for CIS/MS. | 5 years or clinical conversion to MS

CONTACTS AND LOCATIONS:
Overall Officials: Staley A Brod, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas - Houston, Houston, Texas, United States